CLINICAL TRIAL: NCT03573804
Title: The Prone to Supine Breast MRI Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Timothy B. Rooney, MD, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D17168
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Results first posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Locator
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prone to Supine MRI (Experimental): The patient will be placed in the prone position and undergo a standard Gd contrast-enhanced bilateral breast MRI. Immediately after the prone MRI is completed, the patient will be repositioned for the supine MRI. Prior to starting the prone MRI, the study MRI technician/investigator will explain to the patient and practice with the patient the steps needed to transition from the prone to the supine MRI, so as to facilitate a timely transition. Additional MRI images will only take about 10-15 minutes to obtain and will not require a second injection of contrast material.
  Interventions: Other: Prone to Supine MRI

INTERVENTIONS:
Other: Prone to Supine MRI — The patient will be placed in the prone position and undergo a standard Gd contrast-enhanced bilateral breast MRI. Immediately after the prone MRI is completed, the patient will be repositioned for the supine MRI. Prior to starting the prone MRI, the study MRI technician/investigator will explain to the patient and practice with the patient the steps needed to transition from the prone to the supine MRI, so as to facilitate a timely transition. Additional MRI images will only take about 10-15 minutes to obtain and will not require a second injection of contrast material.

SUMMARY:
The purpose of this study is to determine whether a supine MRI obtained immediately after a standard diagnostic prone MRI exam, without a second injection of gadolinium (Gd) contrast material, would be of sufficient quality to allow the Radiologist to define the tumor edges ("segment" the tumor) so that a 3-D image of the tumor can be generated to form a BCL.

DETAILED DESCRIPTION:
The purpose of this study is to find out whether additional MRI images taken with patients in a different position after completing a standard MRI are of sufficient quality to allow a radiologist to identify the edges of the tumor.

These additional MRI images will only take about 10-15 minutes to obtain and will not require a second injection of contrast material.The information gathered in this study will make it more feasible to use a new device called the "breast cancer locator" to help surgeons more accurately remove breast cancers.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Female gender.
* Histologic diagnosis of invasive breast cancer or ductal carcinoma in situ
* Tumor size at least 1 cm in diameter as visualized on mammogram or US.
* A diagnostic breast MRI is considered to be clinically indicated.
* Ability to voluntarily provide informed consent to participate prior to any study-related assessments/procedures being conducted.

Exclusion Criteria:

* Absolute contraindication to MRI, including presence of implanted electrical device (pacemaker or neurostimulator), aneurysm clip, or metallic foreign body in or near eyes.
* Severe claustrophobia.
* Contraindication to use of gadolinium-based intravenous contrast, including life- threatening allergy or compromised renal function (eGFR < 30 ml/min/1.73m2).
* History of median sternotomy.
* Pregnancy. Patient attestation that they are not pregnant will be acceptable.
* Patients who have received neoadjuvant chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Rooney, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barth RJ Jr, Krishnaswamy V, Paulsen KD, Rooney TB, Wells WA, Rizzo E, Angeles CV, Marotti JD, Zuurbier RA, Black CC. A Patient-Specific 3D-Printed Form Accurately Transfers Supine MRI-Derived Tumor Localization Information to Guide Breast-Conserving Surgery. Ann Surg Oncol. 2017 Oct;24(10):2950-2956. doi: 10.1245/s10434-017-5979-z. Epub 2017 Aug 1. PMID 28766199
- [Background] Leong CS, Daniel BL, Herfkens RJ, Birdwell RL, Jeffrey SS, Ikeda DM, Sawyer-Glover AM, Glover GH. Characterization of breast lesion morphology with delayed 3DSSMT: an adjunct to dynamic breast MRI. J Magn Reson Imaging. 2000 Feb;11(2):87-96. doi: 10.1002/(sici)1522-2586(200002)11:23.0.co;2-e. PMID 10713939

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prone to Supine MRI
Started | 72
Completed | 62
Not Completed | 10
Not completed — claustrophobia or MRI table problems | 10

BASELINE CHARACTERISTICS:
Arm/Group | Prone to Supine MRI
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 68
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 71
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Successful Segmentation of Supine MRI Images
Description: Determine what number of cases that can be successfully segmented both from using post-contrast prone MRI images and also from using post contrast supine MRI images.
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Groups:
- Prone to Supine MRI Evaluated by Radiologist A: Radiologist A, number of participants successfully segmented
- Prone to Supine MRI Evaluated by Radiologist B: Radiologist B, number of participants successfully segmented
Arm/Group | Prone to Supine MRI Evaluated by Radiologist A | Prone to Supine MRI Evaluated by Radiologist B
Number analyzed (Participants) | 62 | 62
Participants | 54 | 61

2. Secondary Outcome: Enhancement Quantification, as Measured by Signal Intensity - Segmented Tumor
Description: Compare the signal intensity with that obtained at tumor location on the prone and supine imaging. The amount of enhancement at the tumor site = segmented tumor.
Time Frame: 30 minutes
Population: One participant was not able to complete both the Prone and Supine Imaging and was excluded.
Measure: Mean (Full Range); unit: Tesla per second
Groups:
- Prone Images: Prone MRI images
- Supine Images: Supine MRI images
Arm/Group | Prone Images | Supine Images
Number analyzed (Participants) | 61 | 61
Tesla per second | 370.09 [63.33 to 958.31] | 594.77 [81.50 to 1520.94]
Statistical Analysis 1: Comparison: Prone Images vs Supine Images; Regions of interest (ROIs) for tumor were defined by the radiologist segmentation of tumor in supine and prone positions. ROIs for the surrounding tissue were selected such that tumor and normal regions had equal volumes. The alpha level was assumed to be of 0.05 (dof = 60), and the null hypothesis of equivalence (mu = 0); Test type: Other — A two-tailed paired T-test for equivalence was used to evaluate equivalence between the average raw tumor; p < 0.001, t-test, 2 sided — Using an alpha value of 0.05, dof = 60, the null hypothesis of sample mean equivalence was rejected; A paired two-tailed t-test was used on the paired prone-to-supine tumor intensity values; Mean Difference (Net) = 224.675, 95% CI 2-sided [90.26044 to 359.08956], Standard Error of Mean 67.89

3. Secondary Outcome: Enhancement Quantification, as Measured by Signal Intensity - Tumor Boundary
Description: Compare the signal intensity with that obtained in benign tissue surrounding the tumor on the prone and supine imaging.
Time Frame: 30 minutes
Population: One participant was not able to complete both the Prone and Supine Imaging and was excluded.
Measure: Mean (Full Range); unit: Tesla per second
Arm/Group | Prone Images | Supine Images
Number analyzed (Participants) | 61 | 61
Tesla per second | 217.96 [42.3 to 534.75] | 383.80 [35.53 to 1108.08]
Statistical Analysis 1: Comparison: Prone Images vs Supine Images; Regions of interest (ROIs) for surrounding tissues were selected as the surrounding benign tissue regions directly adjacent to the segmented tumor regions. Tumor and surrounding regions had equal volumes. The mean surrounding region intensities reported were all calculated from the prone and supine T1-weighted MR images segmented by the radiologist; Test type: Other — A two-tailed paired T-test was used to compare sample means in between the prone and supine mean benign tissue intensities; p < 0.001, t-test, 2 sided — Using an alpha value of 0.05, dof = 60, the null hypothesis of sample mean equivalence was rejected; A paired two-tailed t-test was used on the paired prone-to-supine normal tissue intensity values; Mean Difference (Net) = 165.833, 95% CI 2-sided [78.34708 to 253.31892], Standard Error of Mean 44.19

4. Secondary Outcome: Enhancement Quantification- Tumor-to-Background Ratio
Description: Mean MRI signal of the segmented tumor divided by the mean MRI signal of the surrounding tissue which has an equal volume to the tumor. The difference between tumor and benign breast tissue is the tumor-to-background ratio
Time Frame: 30 minutes
Population: One participant was not able to complete both the Prone and Supine Imaging and was excluded.
Measure: Mean (Full Range); unit: Ratio
Arm/Group | Prone Images | Supine Images
Number analyzed (Participants) | 61 | 61
Ratio | 1.74 [1.07 to 3.56] | 1.62 [0.88 to 3.86]
Statistical Analysis 1: Comparison: Prone Images vs Supine Images; The ratios of tumor-to-surrounding tissue intensities, as calculated in Secondary Objective Part A, were compared between prone and supine T1-weighted MR image scans; Test type: Other — A two-tailed paired T-test was used to compare sample means in between the prone and supine tumor-to-surrounding tissue ratios; p = 0.0058, t-test, 2 sided — Using an alpha value of 0.05, dof = 60, the null hypothesis of sample mean equivalence was rejected; A two-tailed paired T-test was used to compare sample means in between the prone and supine tumor-to-surrounding tissue ratios; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.04209 to 0.28209], Standard Error of Mean 0.08

5. Secondary Outcome: Time to Position and Obtain Supine Images
Description: Calculate the additional time needed to obtain supine MRI images. After the completion of Prone imaging, the patient was removed from the MRI, turned over to the supine position, new coils placed, and returned to the MRI for additional imaging. The aggregate time to accomplish these tasks are noted in minutes.
Time Frame: 30 Minutes
Measure: Median (Full Range); unit: minutes
Arm/Group | Prone to Supine MRI
Number analyzed (Participants) | 62
minutes | 7.25 [5.0 to 15.92]

6. Secondary Outcome: Overall Comfort for Prone and Supine Positions
Description: Quantify the perceived comfort level of the prone and supine MRI as reported by participants. A single question using a Likert scale was was used. The scale range was 0 to 5, where 0 = no pain, completely comfortable and 5 = considerable discomfort.
Time Frame: Within 15 minutes of the scan
Population: This assessment of overall perceived comfort was added to the study during the study period, and only the last 28 patients evaluated their overall comfort with the prone and supine portions of the examination.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Overall Comfort - Prone Participants.: Quantify the perceived comfort level of the prone MRI as reported by participants.
- Overall Comfort Participants - Supine: Quantify the perceived comfort level of the supine MRI as reported by participants.
Arm/Group | Overall Comfort - Prone Participants. | Overall Comfort Participants - Supine
Number analyzed (Participants) | 28 | 28
units on a scale | 1.82 [0 to 5] | 0.61 [0 to 5]
Statistical Analysis 1: Comparison: Overall Comfort - Prone Participants. vs Overall Comfort Participants - Supine; Test type: Superiority; p = 0.00049664, Students two-tailed paired t-test

ADVERSE EVENTS:
Time Frame: Two weeks after scans
Arm/Group | Prone to Supine MRI
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT03573804/Prot_SAP_000.pdf